CLINICAL TRIAL: NCT03373227
Title: Phase II, Single-Center, Open-Label Study Evaluating the Comparable Efficacy of Tacrolimus Extended Release Tablets (Envarsus®) to the Standard of Care (SOC) Twice Daily Tacrolimus (Prograf®) Dosing Regimen
Brief Title: Phase II Study Evaluating the Efficacy of Tacrolimus Extended Release Tablets to Twice Daily Tacrolimus Dosing Regimen
Acronym: Veloxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-178
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2023-01

CONDITIONS: Heart Transplant Rejection; Graft Failure; Compliance, Patient
Keywords: Heart Transplant
MeSH Terms: conditions — Patient Compliance | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective (Experimental): 25 adult male or female recipients of a heart transplant will be prospectively enrolled to once-daily therapy with Envarsus tablets. Time of initiation will follow current standard of care.
  Interventions: Drug: Envarsus
- Retrospective (No Intervention): 25 age/gender-matched subjects who are receiving twice daily dosing with Prograf will be identified from the transplant center database and contacted to be consented, after which their results will be analyzed retrospectively.

INTERVENTIONS:
Drug: Envarsus — Patients will take once daily Envarsus
  Arms: Prospective

SUMMARY:
This phase II, single-center, open-label study will evaluate the comparable efficacy of tacrolimus extended release tablets (Envarsus®) to the standard of care (SOC) twice daily tacrolimus (Prograf®) dosing regimen post-cardiac transplantation.

DETAILED DESCRIPTION:
This is a prospective, open-label, 2-arm, clinical trial to evaluate the efficacy of extended release tacrolimus (Envarsus) once-daily in comparison to Prograf capsules twice-daily after heart transplantation receiving the standard of care twice daily dosing with tacrolimus (Prograf).

Secondary objectives are to compare the compliance, safety and efficacy of once a day dosing (Envarsus) versus twice a day dosing (Prograf) and to evaluate the short term safety and tolerability of Envarsus.

Approximately 25 adult male or female recipients of a heart transplant will be prospectively enrolled to once-daily therapy with Envarsus tablets. Time of initiation will follow current standard of care. In addition, 25 age/gender-matched subjects who are receiving twice daily dosing with Prograf will be identified from the transplant center database and contacted to be consented, after which their results will be analyzed retrospectively.

The Termination Visit will occur on Day 182 (± 2 days) for subjects who complete the study treatment. Subjects who receive the first dose of study drug but withdraw from the study or terminate study treatment for any reason should complete all the procedures outlined for the Termination Visit.

The follow-up safety assessment may be conducted via telephone or at a study visit if needed for clinical follow-up on any safety issues). The follow-up safety assessment is to take place approximately 30 days (±5 days) after the last administration of study treatment, whether the subject completed study treatment or withdrew or terminated treatment early.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age
* Able to comply with medication regimen
* Subjects must have the capacity to understand and sign the informed consent form
* Heart-only transplant recipients

Exclusion Criteria:

* Subject currently enrolled in another interventional research trial
* History of hypersensitivity/adverse reaction to tacrolimus
* Patient taking Rapamycin (sirolimus) or cyclosporine (Neoral/Gengraf)
* Simultaneous multiple organ transplant recipients
* Liver transplant recipients / candidates

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Rejection and Graft Failure | 2 years
  Evaluate effect on rejection and graft failure by comparing adverse events in standard of care versus experimental groups

SECONDARY OUTCOMES:
Effect of Compliance on Rejection and Graft Failure | 2 years
  To compare complications that lead to acute rejection and graft failure based on patient compliance to once a day dosing versus twice a day dosing

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Hall, MD, FACC, FHFSA, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No